CLINICAL TRIAL: NCT05074550
Title: Phase I, Open-Label, Multicentre, Dose-Escalation Study to Evaluate the Safety and Pharmacokinetics of A Single Intravenous PPMX-T003 in Polycythemia Vera
Brief Title: Safety Evaluation Study for Patients With Polycythemia Vera
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Perseus Proteomics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PPMX-T003-CT102
Record Dates: First submitted 2021-09-14; First posted 2021-10-12 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2022-11

CONDITIONS: Polycythemia Vera
Keywords: Myeloproliferative neoplasms
MeSH Terms: conditions — Polycythemia Vera; Myeloproliferative Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PPMX-T003 (Experimental): This drug should be administered within 48 hours after the phlebotomy. In addition, as a dose escalation design, 4 doses of 0.25 mg/kg, 0.4 mg/kg, 0.64 mg/kg, and 1 mg/kg are administered to the same subject, when the next phlebotomy required during observation period after the 1st administration.
  Interventions: Drug: PPMX-T003

INTERVENTIONS:
Drug: PPMX-T003 — As an observation and evaluation method, for each dose, in principle, inpatient observation is performed for 1 week from the day before administration, and then safety and pharmacodynamic tests are evaluated by visiting the hospital every 2 weeks.

SUMMARY:
This is PhaseI Dose-Escalation Study to Evaluate the Safety and Pharmacokinetics of PPMX-T003 in Polycythemia Vera

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PV according to either the 2008 or 2016 WHO classification criteria
* PV patients being only treated with phlebotomy and the interval is 4-9 weeks

Exclusion Criteria:

* Patients administrated drugs for PV treatment such as hydroxyurea or ruxolitinib (aspirin is excluded)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Patients Experiencing Treatment-emergent Adverse Events (TEAEs) in the Study | 45 weeks

SECONDARY OUTCOMES:
Evaluation of pharmacokinetics of PPMX-T003 after single dose | Day1,Day2,Day7
  Observed maximum plasma concentration [Cmax]
Evaluation of pharmacokinetics of PPMX-T003 after single dose | Day1,Day2,Day7
  Terminal elimination rate constant [λz]
Evaluation of pharmacokinetics of PPMX-T003 after single dose | Day1,Day2,Day7
  Area under the concentration-time curve from pre-dose [time 0] to the time of the last quantifiable concentration [AUC0-t]
Evaluation of pharmacokinetics of PPMX-T003 after single dose | Day1,Day2,Day7
  Area under the concentration-time curve from pre-dose [time 0] extrapolated to infinite time [AUC0-inf]
Evaluation of pharmacokinetics of PPMX-T003 after single dose | Day1,Day2,Day7
  Apparent terminal half-life [t½]
Evaluation of pharmacokinetics of PPMX-T003 after single dose | Day1,Day2,Day7
  Apparent systemic clearance [CL]
Evaluation of pharmacokinetics of PPMX-T003 after single dose | Day1,Day2,Day7
  Volume of distribution [Vd]
Examining the expression rate of anti-drug antibodies (ADA) | Day1,Day21,up to 45weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Shimane University Hospital, Izumo, Shimane
  - Osaka City University Hospital, Osaka

REFERENCES:
- [Derived] Gorak EJ, Otterstatter M, Al Baghdadi T, Gillis N, Foran JM, Liu JJ, Bejar R, Gore SD, Kroft SH, Harrington A, Saber W, Starczynowski D, Rollison DE, Zhang L, Moscinski L, Wilson S, Thompson J, Borchert C, Sherman S, Hebert D, Walker ME, Padron E, DeZern AE, Sekeres MA. Discordant pathologic diagnoses of myelodysplastic neoplasms and their implications for registries and therapies. Blood Adv. 2023 Oct 24;7(20):6120-6129. doi: 10.1182/bloodadvances.2023010061. PMID 37552083